CLINICAL TRIAL: NCT02309190
Title: Transpulmonary Pressures in Mechanical Ventilated Patients With Morbid Obesity
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Rosa Estrada Y Martin, Associate Professor, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-14-0444
Record Dates: First submitted 2014-09-16; First posted 2014-12-05 (Estimated); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Mechanical Ventilation Complication; Respiratory Insufficiency
Keywords: Transpulmonary pressure - morbid obesity
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- transpulmonary pressures: Esophageal balloon to measure transpulmonary pressures. PEEP adjustment as per transpulmonary pressures.

SUMMARY:
The study consists in determine the transpulmonary pressure in morbidly obesity patients that require mechanical ventilation.

* both gender
* only adults
* Medical intensive care patients.

DETAILED DESCRIPTION:
We are studying adult patients with morbid obesity with respiratory failure requiring mechanical ventilation.

We are measuring transesophageal presssures to estimate ideal PEEP and evaluate hemodynamic parameters.

ELIGIBILITY:
Inclusion Criteria:

* both gender
* morbid obesity
* hemodynamically stable

Exclusion Criteria:

* pregnant patients
* cirrhotic patients with esophageal varicose

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults mechanically ventilated with morbid obesity
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Transpulmonary pressure | one year
  We will record the changes in transpulmonary pressure after adjusting PEEP (measure in cmH2O).

SECONDARY OUTCOMES:
hemodynamics | one year
  we will review hemodynamic changes while adjusting PEEP (BP, HR).

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Texas - HSC at Houston, Houston, Texas, United States